CLINICAL TRIAL: NCT06789250
Title: Co-occurence of Mental Illness and Problematic Alcohol Use: an Internet-based Cognitive Behavior Therapy Intervention
Acronym: CoMiT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CoMiT
Record Dates: First submitted 2024-12-18; First posted 2025-01-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Drinking Related Problems; Alcohol Use Disorders; Depressive Disorders; Mental Illness; Mental Stress; Mental and Behavioral Disorders; Sleep Problems; Stress Disorders; Anxiety Disorder/Anxiety State
Keywords: Internet intervention; Depression; Anxiety; Individually tailored; Transdiagnostic; Internet-based cognitive behavioral therapy (ICBT); Stress; Sleeping disorders; Mental illness; Harmful alcohol use; Alcohol addiction
MeSH Terms: conditions — Alcoholism; Depressive Disorder; Mental Disorders; Stress, Psychological; Parasomnias; Stress Disorders, Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): 10 weeks of therapist supported, individually tailored, internet-based cognitive behavior therapy with weekly and on-demand support by a therapist.
  Interventions: Behavioral: Internet-based cognitive behavior therapy
- Control group (No Intervention): A wait-list control condition where the participants recieve weekly attention from the research team therapists. After the treatment group has finished their 10 weeks of treatment and post-treatment measures has been collected, the control group receive the same treatment program as the treatment group.

INTERVENTIONS:
Behavioral: Internet-based cognitive behavior therapy — The intervention within this study is based on cognitive behavioral therapy principles and adapted to target harmful alcohol use and mild to moderate alcohol use disorder co-occuring with psychological symptoms of depression, anxiety, stress and/or sleeping disorder. The 10 weeks of individually tailored treatment include psycho-educational texts as well as examples and exercises supported by a therapist.
  Arms: Treatment group

SUMMARY:
The goal of this clinical trial is to learn if internet-based cognitive behavior therapy (ICBT ) works to treat co-occurent of problematic alcohol use and mental illness including mild to moderate symptoms of either depression, anxiety, stress or disturbed sleep.

The main questions the study aims to answer are:

* Does the ICBT program lower the self-rated suffering from mental illness?
* Does the ICBT program lower the self-reported alcohol intake? Researchers will compare the ICBT program to the participants who are rancomized to a control grout that receives weekly attention from the research team, to see if the treatment works. In both groups, the participants will have the opportunity to ask for support from a therapist during the week days.

Participants are adults living in Sweden. They will:

* Receive an ICBT program supported by a trained therapist. It consists of modules that the participants will work with on their computer for 10 weeks. Some modules will be compulsory and other optional for the participants.
* Fill out forms to rate their mental illness and alcohol intake at the start and the end of the study as well as once every week during treatment.

Primary outcome measures are depression, anxiety and stress symptoms (measured with Depression Anxiety and Stress Scale 21 (DASS-21)) and alcohol intake measured with self-reported amounts. Other, secondary, outcome measures used will for example be about insomnia symptoms and disability assessment. Pre-treatment measurement, post-treatment measurement and 6-months and 12-months follow up is planned to be collected through an online survey.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* AUDIT ≥ 6 points for women and ≥ 8 points for men
* Symptoms of depression, anxiety disorder and/or stress-related illness
* Adequate ability to speak, read and write Swedish
* Having access to the internet and a smartphone, computer or other device.

Exclusion Criteria:

* Ongoing psychological treatment.
* Ongoing medication for AUD
* Recent changes (within the past three months) in psychiatric medication or planned changes during the treatment period. New medication prescribed during the study shall be reported but will not lead to exclusion
* Severe psychiatric disorders based on a Mini-International Neuropsychiatric Interview (MINI) interview and reported medical history
* Severe medical conditions that may impede participation in the study
* Severe cognitive impairment
* Current suicidality
* Severe alcohol addiction where specialized treatment is more appropriate
* Risk for severe alcohol withdrawal symptoms with a need for medical treatment. Participation is possible after completing alcohol withdrawal treatment within the ordinary health-care system, accessible to the Swedish population.
* Substance use disorder, other than alcohol or nicotine, within the past six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
High-risk alcohol drinking days (HDD) | Change between baseline and end of treatment (expected 3 months after baseline). Additionally the change between baseline and 6 months and 12 months follow-up after end of treatment (hence expected 9 months and 15 months after baseline).
  Amount of alcohol use measured in number of high-risk drinking days (HDD), defined according to the World Health Organization (WHO) risk drinking levels, as a daily intake of ≥60 grams pure alcohol for men and ≥40 g for women. Alcohol intake is assessed by self-reported number of standard glasses of alcohol beverage (each containing 12 g of pure ethanol). This is self-reported each day with Timeline Follow Back (TLFB) procedure and then converted to grams pure alcohol.
The Depression Anxiety Stress Scales (DASS-21) | Change between baseline and end of treatment (expected 3 months after baseline). Additionally the change between baseline and 6 months and 12 months follow-up after end of treatment (hence expected 9 months and 15 months after baseline).
  Measure of self-reported symptoms of depression, anxiety and stress. Consists of 21 items that are scored on a range between 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). Scores can range between 0 and 63 points. Higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Number of self-reported alcohol abstinent days | At baseline, every 7 days during treatment, at end of treatment (expected 3 months after baseline) and 6 months and 12 months after end of treatment (expected 9 months and 15 months after baseline).
  Measure of number of self-reported alcohol abstinent days. Alcohol intake is assessed by self-reported number of standard glasses of alcohol beverage. This is self-reported each day with Timeline Follow Back (TLFB) procedure. A day with zero reported alcohol use is considered an abstinent day.
Total amount of alcohol intake | At baseline, every 7 days during treatment, at end of treatment (expected 3 months after baseline) and 6 months and 12 months after end of treatment (expected 9 months and 15 months after baseline).
  Measure of self-reported alcohol intake. Alcohol intake is assessed by self-reported number of standard glasses of alcohol beverage (each containing 12 g of ethanol). This is self-reported each day with Timeline Follow Back (TLFB) procedure covering the last 7 days and then converted to grams of ethanol.
Alcohol craving Visual analogue scale (AC-VAS) | At baseline, every 7 days during treatment, at end of treatment (expected 3 months after baseline) and 6 months and 12 months after end of treatment (expected 9 months and 15 months after baseline).
  Measure of perceived alcohol craving by self-rating on a visual analogue scale (VAS) ranging from 0 to 100 where 0 denotes no craving and 100 the worst possible craving.
Insomnia Severity Index (ISI) | At baseline, at end of treatment (expected 3 months after baseline) and follow-up 6 months and 12 months after end of treatment (expected 9 months and 15 months after baseline).
  Measure of insomnia and sleep related-difficulties that consists of seven items. Higher self-reported scores indicate greater sleep related-difficulties. Scores can range from 0 to 28.
Perceived Stress Scale (PSS-10) | At baseline, at end of treatment (expected 3 months after baseline) and follow-up 6 months and 12 months after end of treatment (expected 9 months and 15 months after baseline).
  A self-report questionnaire that measures perceived stress, sense of control and self-efficacy. It contains 10 items that are scored on a range between 0 (never) to 4 (very often). The total score range is between 0-40 and a higher score reflects higher levels of perceived stress.
The World Health Organization Disability Assessment Schedule (WHODAS-12) | At baseline, at end of treatment (expected 3 months after baseline) and follow-up 6 months and 12 months after end of treatment (expected 9 months and 15 months after baseline).
  A self-report questionnaire that measures disability due to health conditions. It contains 12 items that are scored on a range between 0 (none) to 4 (extreme). The total score ranges between 0 to 48 and a higher score reflects a higher degree of disability.
The Short Index of Problems (SIP) | At baseline, at end of treatment (expected 3 months after baseline) and follow-up 6 months and 12 months after end of treatment (expected 9 months and 15 months after baseline).
  A self-report questionnaire for measuring drinking consequences in problem drinkers during the last 3 months. It contains 15 items that are scored on a range between 0 (never) to 3 (daily). The total score ranges between 0 to 45 and a higher score reflects more negative consequences from alcohol intake.
Montgomery-Åsberg Depression Rating Scale (MADRS) | At baseline, at mid-treatment (expected 6 weeks after baseline), at end of treatment (expected 3 months after baseline) and follow-up at 6 months and 12 months after end of treatment (expected 9 months and 15 months after baseline).
  A self-report questionnaire that measures symptoms of depression and detects signs of increased suicidality. It contains 9 items that are scored on a range between 0 (none) to 6 (extreme). The total score ranges between 0 to 54 and a higher score reflects more symptoms of depression.
Alcohol Use Disorder Identification Test | At baseline, at end of treatment (expected 3 months after baseline) and follow-up 6 months and 12 months after end of treatment (expected 9 months and 15 months after baseline).
  A self-report questionnaire to assess alcohol consumption, drinking behaviors, and alcohol-related problems. 10 items and scores ranging from 0-40 with higher scores indicating a higher level of problematic alcohol use.
B-Phosphatidylethanol (PEth) | At baseline and at end of treatment (expected 3 months after baseline).
  A biomarker of alcohol intake sampled with a measure called dried blood spot (DBS), that the participant can sample at home. Measures amount of Phosphatidylethanol (µmol/l) in blood,

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Professor, Principal Investigator — Linkoeping University
Locations (2):
- Sweden (2):
  - Linköping University, Linköping
  - Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County

REFERENCES:
- See also: Homepage for information and registration for participation — http://www.comitstudien.se